CLINICAL TRIAL: NCT02908295
Title: Rectal Misoprostol in Women Undergoing Myomectomy for Intraoperative Blood Loss: A Randomized Placebo-controlled Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RJMISO
Record Dates: First submitted 2016-09-16; First posted 2016-09-20 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2016-09

CONDITIONS: Misoprostol, Blood Loss, Myomectomy
MeSH Terms: conditions — Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Rectal Misoprostol Misoprostol 400 mcg (200 mcg/tablet) or 2 tablets were given rectally at 15 - 30 minutes prior the operation
  Interventions: Drug: Rectal Misoprostol
- B (Placebo Comparator): Rectal Vitamin B6 Vitamin B6 (Placebo) 200 mg (100 mg/tablet) or 2 tablets were given rectally at 15 - 30 minutes prior the operation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rectal Misoprostol — Rectal Misoprostol Misoprostol 400 mcg (200 mcg/tablet) or 2 tablets were given rectally at 15 - 30 minutes prior the operation
  Other Names: Cytotec
  Arms: A
Drug: Placebo — Rectal Vitamin B6 Vitamin B6 (Placebo) 200 mg (100 mg/tablet) or 2 tablets were given rectally at 15 - 30 minutes prior the operation
  Other Names: Besix
  Arms: B

SUMMARY:
Comparison of efficacy of rectal misoprostol for reduction amount of blood loss in women undergoing myomectomy, both open and laparoscopic approach

DETAILED DESCRIPTION:
According to development of reproductive technology to assist infertile women, rate of myomectomy increases. During this operation, surgeons would deal with hypervascular masses with raw surfaces that tend to bleeding. Interventions to diminish bleeding were studied such as using misoprostol, vasopressin, transamenic acid along with mechanical intervention such as tourniquet and uterine artery ligation. But in Rajavithi hospital, such procedures aren't generally used because of fewer cases and also lacks of supporting data. Misoprostol, used in gynecologic patients for a long time with a wide safety margin acts at prostaglandin receptors of myometrium to stimulate contraction that constricts uterine vessels that lead to decreasing amount of bleeding during the operation. This led to the experimental study of rectal misoprostol administered at 15 - 30 minutes prior the operation to decrease blood loss and also blood transfusion rates. Our study also gather data about adverse effect that subject experienced after drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Patient provisionally diagnosed with leiomyoma of uterus with less than 10 cm diameter
* Patient undergoing myomectomy, both open and laparoscopic approach
* Patient aged 25 - 50 years
* Patient able to give free and informed consent and who agrees to participate bu signing the consent form
* Patient able to speak and understand Thai
* Patient able to complete the questionnaire

Exclusion Criteria:

* Patient who was pathologically diagnosed apart from leiomyoma
* Patient with leiomyoma FIGO type 0
* Patient who has medical conditions that increase bleeding tendency, such as thrombocytopenia, coagulopathy, renal insufficiency, uncontrolled diabetes mellitus, taking antiplatelets or anticoagulants less than 7 days prior the surgery
* Patient who takes prostaglandin analogs and/or antagonists (NSAIDS) less than 7 days prior the surgery.
* Patient who may take higher risks of misoprostol adverse effect such as hypertension, ischemic heart disease, glaucoma, asthma
* Patient who had and allergic reaction to misoprostol or vitamin B6

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Mean intraoperative blood loss in both groups | Within 3 hours

SECONDARY OUTCOMES:
Mean difference of hemoglobin | within 24 hours
Incidence of blood transfusion | within 72 hours
Incidence of unplanned operation | within 72 hours
Incidence of adverse events | within 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No